CLINICAL TRIAL: NCT02951312
Title: Single-dose, Dose Escalation Study to Assess the Safety, Tolerability, Pharmacokinetics and Bronchodilatory Effects of Glycopyrrolate Inhalation Solution (GIS) Using a High Efficiency Nebulizer in Patients With COPD
Brief Title: Assessment of the Safety and Ability of a Once-a-day Dose of an Orally Inhaled Medicine [ie, Glycopyrrolate Inhalation Solution = GIS] to Improve Airflow in the Lungs When Delivered With an Electronic eFlow Nebulizer System in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sunovion Respiratory Development Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EP-101-01; 2009-010821-38 (EudraCT Number)
Record Dates: First submitted 2016-10-26; First posted 2016-11-01 (Estimated); Results first posted 2018-04-30 (Actual); Last update posted 2018-04-30 (Actual); Status verified 2018-03

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Emphysema; Chronic bronchitis; COPD; Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Emphysema; Bronchitis, Chronic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (7):
- Glycopyrrolate Inhalation Solution 25mg (Experimental): Glycopyrrolate Inhalation Solution 25 μg via eFlow nebulizer, once daily
  Interventions: Drug: Glycopyrrolate Inhalation Solution 25mg
- Glycopyrrolate Inhalation Solution 75mg (Experimental): Glycopyrrolate Inhalation Solution 75 μg via eFlow nebulizer, once daily
  Interventions: Drug: Glycopyrrolate Inhalation Solution 75mg
- Glycopyrrolate Inhalation Solution 200mg (Experimental): Glycopyrrolate Inhalation Solution 200 μg via eFlow nebulizer, once daily
  Interventions: Drug: Glycopyrrolate Inhalation Solution 200mg
- Glycopyrrolate Inhalation Solution 200mg Jet (Experimental): Glycopyrrolate Inhalation Solution 200 μg via jet nebulizer, once daily
  Interventions: Drug: Glycopyrrolate Inhalation Solution 200mg Jet
- Glycopyrrolate Inhalation Solution 500mg (Experimental): Glycopyrrolate Inhalation Solution 500 μg via eFlow nebulizer, once daily
  Interventions: Drug: Glycopyrrolate Inhalation Solution 500mg
- Glycopyrrolate Inhalation Solution1000mg (Experimental): Glycopyrrolate Inhalation Solution 1000 μg via eFlow nebulizer, once daily
  Interventions: Drug: Glycopyrrolate Inhalation Solution1000mg
- Placebo 0.5 mL (Placebo Comparator): Placebo 0.5 mL via jet nebulizer, once daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Glycopyrrolate Inhalation Solution 25mg — 25 μg oral inhalation via eFlow Nebulizer, once daily
  Other Names: GIS
  Arms: Glycopyrrolate Inhalation Solution 25mg
Drug: Glycopyrrolate Inhalation Solution 75mg — 75 μg oral inhalation via eFlow Nebulizer, once daily
  Other Names: GIS
  Arms: Glycopyrrolate Inhalation Solution 75mg
Drug: Glycopyrrolate Inhalation Solution 200mg — 200 μg oral inhalation via eFlow Nebulizer, once daily
  Other Names: GIS
  Arms: Glycopyrrolate Inhalation Solution 200mg
Drug: Glycopyrrolate Inhalation Solution 200mg Jet — 200 μg oral inhalation via inhalation via jet nebulizer, once daily
  Other Names: GIS
  Arms: Glycopyrrolate Inhalation Solution 200mg Jet
Drug: Glycopyrrolate Inhalation Solution 500mg — 500 μg oral inhalation via eFlow nebulizer, once daily
  Other Names: GIS
  Arms: Glycopyrrolate Inhalation Solution 500mg
Drug: Glycopyrrolate Inhalation Solution1000mg — 1000 μg oral inhalation via eFlow nebulizer, once daily
  Other Names: GIS
  Arms: Glycopyrrolate Inhalation Solution1000mg
Drug: Placebo — Placebo 0.5 mL oral inhalation via jet nebulizer, once daily
  Arms: Placebo 0.5 mL

SUMMARY:
The study assessed the safety and ability of several doses of an orally inhaled medicine [ie, Glycopyrrolate Inhalation Solution = GIS] to improve airflow in the lungs when delivered with an electronic eFlow nebulizer system in patients with Chronic Obstructive Pulmonary Disease (COPD). The study was conducted in 12 patients in 2 parts. Part 1 was designed to find the once-a- day GIS dose that produced the highest improvement in lung airflow. Part 2 tested the GIS dose with the highest improvement in lung airflow and a placebo (ie, no drug) delivered by a general purpose nebulizer. The airflow improvements of the same GIS dose were compared between the two nebulizer systems to determine what effect the device had on GIS delivery.

DETAILED DESCRIPTION:
In Part I, 12 subjects were randomly allocated to one of 2 cohorts, running in parallel. The 6 cohort 1 subjects received 25 mg and then 200 mg during their treatment periods 1 and 2, respectively. The 6 cohort 2 subjects received 75mg, 500mg, and 1000 mg during their treatment periods 1, 2, and 3, respectively. During Part II of the study, the same 12 subjects from Part I were randomized to receive either 200 mg jet or placebo in a 1:1 ratio.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients aged 40 through 75 years, inclusive
2. A clinical diagnosis of COPD according to the GOLD guidelines
3. Current smokers or ex-smokers with at least 10 pack-year smoking history (e.g., at least 1 pack/day for 10 years, or 10 packs/day for 1 year)
4. Post-bronchodilator FEV1 40-80% of predicted normal
5. Post-bronchodilator FEV1/FVC ratio < 0.70
6. Improvement in FEV1 >12% (minimum 150 mL) following inhalation of ipratropium bromide
7. Ability to perform reproducible spirometry according to the ATS/ERS guidelines
8. If female and of childbearing potential, must have had a negative pregnancy test and was not lactating at the Screening Visit, and was using one of the following acceptable means of birth control throughout the study:

   * Post-menopausal for at least two years
   * Surgically sterile
   * Oral contraceptives (taken for at least one month prior to the Screening Visit)
   * Approved implantable or injectable contraceptives (e.g., Norplant®, Depo-Provera® or equivalent)
   * Barrier methods (e.g., condoms with spermicide)
   * Intrauterine device (i.e., IUD)
   * Vasectomy of male partner
   * Non-heterosexual life style
9. Willing and able to provide written informed consent

Exclusion Criteria:

1. Current evidence or recent history of any clinically significant disease (other than COPD) or abnormality in the opinion of the Investigator that would put the patients at risk or which would compromise the quality of the study data; including but not limited to cardiovascular disease, myocardial infraction, hypertension, arrhythmia, diabetes, neurological or neuromuscular disease, liver disease, gastrointestinal disease or electrolyte abnormalities.
2. Recent history of an exacerbation of airway disease within 3 months or need for increased treatments for COPD within 6 weeks prior to the Screening Visit.
3. Regular use of daily oxygen therapy.
4. Use of systemic (e.g., intramuscular or intravenous) steroids within 3 months prior to the Screening Visit
5. Respiratory tract infection within 6 weeks prior to the Screening Visit
6. History of tuberculosis, bronchiectasis or other non-specific pulmonary disease
7. History of urinary retention or bladder neck obstruction type symptoms
8. History of narrow-angle glaucoma
9. Current or recent history (previous 12 months) of excessive use or abuse of alcohol
10. Current evidence or history of abusing legal drugs or the use of illegal drugs or substances
11. History of hypersensitivity or intolerance to aerosol medications
12. Participation in another investigational drug study where drug was received within 30 days prior to the Screening Visit

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2009-05; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ahmet Tutuncu, MD, PhD, Study Chair — Elevation Pharmaceuticals, Inc.(now known as Sunovion Respiratory Development Inc.)

RESULTS

PARTICIPANT FLOW:
Groups:
- 25mg Glycopyrrolate, 200mg Gloycopyrrolate: subjects received 25mg Glycopyrrolate then 200mg Glycopyrrolate in part 1- in part 2 subjects from this group either received 200mg Glycopyrrolate or placebo
- 75mg Glycopyrrolate,500mg Glycopyrrolate,1000mg Glycopyrrolate: subjects received 75mg Glycoprrolate, then, 500mg Glycopyrrolate, then 1000mg Glycopyrrolate in part 1 - in part 2 subjects from this group received either 200mg Glycopyrrolate or placebo
- 200mg Glycopyrrolate Jet: subjects received 200mg Glycopyrrolate
- Placebo: Subjects received placebo
Period: Study Part 1
Arm/Group | 25mg Glycopyrrolate, 200mg Gloycopyrrolate | 75mg Glycopyrrolate,500mg Glycopyrrolate,1000mg Glycopyrrolate | 200mg Glycopyrrolate Jet | Placebo
Started | 6 | 6 | 0 | 0
Completed | 6 | 6 | 0 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Study Part 2
Arm/Group | 25mg Glycopyrrolate, 200mg Gloycopyrrolate | 75mg Glycopyrrolate,500mg Glycopyrrolate,1000mg Glycopyrrolate | 200mg Glycopyrrolate Jet | Placebo
Started | 0 | 0 | 6 | 6
Completed | 0 | 0 | 6 | 6
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants in study
Groups:
- Total: Total of all reporting groups
Arm/Group | 25mg Glycopyrrolate, 200mg Gloycopyrrolate | 75mg Glycopyrrolate,500mg Glycopyrrolate,1000mg Glycopyrrolate | 200mg Glycopyrrolate Jet | Placebo | Total
Number analyzed (Participants) | 6 | 6 | 0 | 0 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 |  |  | 0
  Between 18 and 65 years | 2 | 3 |  |  | 5
  >=65 years | 4 | 3 |  |  | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.2 (3.82) | 63.5 (8.89) |  |  | 41.67 (58.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 |  |  | 5
  Male | 3 | 4 |  |  | 7
Region of Enrollment [Number; unit: participants]
  United Kingdom | 6 | 6 |  |  | 12

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Who Died
Time Frame: 0-47 days
Population: all subjects who received at least one dose of study medication were included in the safety analysis.. A subject received more than one treatment type throughout the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Glycopyrrolate Inhalation Solution 25mg | Glycopyrrolate Inhalation Solution 75mg | Glycopyrrolate Inhalation Solution 200mg | Glycopyrrolate Inhalation Solution 200mg Jet | Glycopyrrolate Inhalation Solution 500mg | Glycopyrrolate Inhalation Solution1000mg | Placebo 0.5 mL
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Subjects With Treatment Emergent SAEs
Description: AEs are defined as existing conditions which worsen or events which occur during the course of the clinical trial after treatment.AEs are defined as existing conditions which worsen or events which occur during the course of the clinical trial after treatment. SAEs are AEs that result in the following outcomes: death, are life-threatening, persistent or significant disability/incapacity, congenital anomaly/birth defect, or important medical events that may have been considered a SAE when, based upon appropriate medical judgment, they may have jeopardized the subject and may have required medical or surgical intervention to prevent one of the outcomes listed in the definition.
Time Frame: 0-47 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Glycopyrrolate Inhalation Solution 25mg | Glycopyrrolate Inhalation Solution 75mg | Glycopyrrolate Inhalation Solution 200mg | Glycopyrrolate Inhalation Solution 200mg Jet | Glycopyrrolate Inhalation Solution 500mg | Glycopyrrolate Inhalation Solution1000mg | Placebo 0.5 mL
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Number of Subjects Who Discontinued Due to AE
Description: AEs are defined as existing conditions which worsen or events which occur during the course of the clinical trial after treatment.
Time Frame: 0-47 days
Population: all subjects who received at least one dose of study medication were included in the safety analysis. . A subject received more than one treatment type throughout the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Glycopyrrolate Inhalation Solution 25mg | Glycopyrrolate Inhalation Solution 75mg | Glycopyrrolate Inhalation Solution 200mg | Glycopyrrolate Inhalation Solution 200mg Jet | Glycopyrrolate Inhalation Solution 500mg | Glycopyrrolate Inhalation Solution1000mg | Placebo 0.5 mL
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Percentage of Subjects With Treatment Emergent AEs
Description: as for outcome 3
Time Frame: 0-47 days
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Glycopyrrolate Inhalation Solution 25mg | Glycopyrrolate Inhalation Solution 75mg | Glycopyrrolate Inhalation Solution 200mg | Glycopyrrolate Inhalation Solution 200mg Jet | Glycopyrrolate Inhalation Solution 500mg | Glycopyrrolate Inhalation Solution1000mg | Placebo 0.5 mL
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6
percentage of participants | 33.3 | 33.3 | 66.7 | 33.3 | 0.0 | 33.3 | 16.7

5. Primary Outcome: Number of Subjects With Clinically Significant Abnormal Vital Signs Reported During the Study
Description: Vital signs were measured at screening, during the study (pre-dose, and 30 and 60 minutes and 2, 4, 8, 12, 24 and 30 hours post-dose) and at post study assessment. The clinical significance of each out of normal range vital sign parameter was determined by the investigator during the study.
Time Frame: 30 hrs post dose
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Glycopyrrolate Inhalation Solution 25mg | Glycopyrrolate Inhalation Solution 75mg | Glycopyrrolate Inhalation Solution 200mg | Glycopyrrolate Inhalation Solution 200mg Jet | Glycopyrrolate Inhalation Solution 500mg | Glycopyrrolate Inhalation Solution1000mg | Placebo 0.5 mL
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0

6. Primary Outcome: Number of Subjects With Clinically Significant Abnormal Laboratory Results Reported During the Study
Description: Clinical safety lab parameters were collected at screening and at the post study follow-up assessment. The clinical significance of each out of normal range laboratory parameter was determined by the investigator during the study.
Time Frame: day 47 (post studyfollow-up assessment)
Population: all subjects who received at least one dose of study medication were included in the safety analysis. A subject received more than one treatment type throughout the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Glycopyrrolate Inhalation Solution 25mg | Glycopyrrolate Inhalation Solution 75mg | Glycopyrrolate Inhalation Solution 200mg | Glycopyrrolate Inhalation Solution 200mg Jet | Glycopyrrolate Inhalation Solution 500mg | Glycopyrrolate Inhalation Solution1000mg | Placebo 0.5 mL
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0

7. Primary Outcome: Number of Subjects With Clinically Significant ECG Parameters Reported During the Study
Description: ECGs were measured at screening, during the study (pre-dose, and 30 and 60 minutes and 2, 4, 8, 12, 24 and 30 hours post-dose) and at post study follow-up assessment.
Time Frame: 30hr post dose
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Glycopyrrolate Inhalation Solution 25mg | Glycopyrrolate Inhalation Solution 75mg | Glycopyrrolate Inhalation Solution 200mg | Glycopyrrolate Inhalation Solution 200mg Jet | Glycopyrrolate Inhalation Solution 500mg | Glycopyrrolate Inhalation Solution1000mg | Placebo 0.5 mL
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0

8. Primary Outcome: Number of Subjects With Clinically Significant Abnormal Laboratory Results Reported During the Study
Description: as for outcome 6
Time Frame: post study follow-up assessment (Day 47)
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Glycopyrrolate Inhalation Solution 25mg | Glycopyrrolate Inhalation Solution 75mg | Glycopyrrolate Inhalation Solution 200mg | Glycopyrrolate Inhalation Solution 200mg Jet | Glycopyrrolate Inhalation Solution 500mg | Glycopyrrolate Inhalation Solution1000mg | Placebo 0.5 mL
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0

9. Primary Outcome: Number of Subjects With Treatment Emergent AEs
Description: AEs are defined as existing conditions which worsen or events which occur during the course of the clinical trial after treatment. SAEs are AEs that result in the following outcomes: death, are life-threatening, persistent or significant disability/incapacity, congenital anomaly/birth defect, or important medical events that may have been considered a SAE when, based upon appropriate medical judgment, they may have jeopardized the subject and may have required medical or surgical intervention to prevent one of the outcomes listed in the definition.
Time Frame: 0-47 days
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Glycopyrrolate Inhalation Solution 25mg | Glycopyrrolate Inhalation Solution 75mg | Glycopyrrolate Inhalation Solution 200mg | Glycopyrrolate Inhalation Solution 200mg Jet | Glycopyrrolate Inhalation Solution 500mg | Glycopyrrolate Inhalation Solution1000mg | Placebo 0.5 mL
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6
Participants | 2 | 2 | 4 | 2 | 0 | 2 | 1

10. Secondary Outcome: Trough FEV1 (Change From Baseline)
Description: Spirometry measurements were conducted in accordance with the current ATS/ERS 2005 guidelines. Trough FEV1 was defined as the spirometry value collected at 24 hours post dose within each Treatment Period.
Time Frame: 24hr post dose
Population: All subjects who received at least one dose of study medication and have at least one post baseline efficacy measurement were included in the efficacy population. A subject received more than one treatment type throughout the study.
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Glycopyrrolate Inhalation Solution 25mg | Glycopyrrolate Inhalation Solution 75mg | Glycopyrrolate Inhalation Solution 200mg | Glycopyrrolate Inhalation Solution 200mg Jet | Glycopyrrolate Inhalation Solution 500mg | Glycopyrrolate Inhalation Solution1000mg | Placebo 0.5 mL
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6
liters | 0.038 (0.157) | 0.087 (0.062) | 0.138 (0.079) | -0.013 (0.098) | -0.017 (0.168) | 0.065 (0.072) | -0.030 (0.070)

11. Secondary Outcome: Peak FEV1 (Percent Change)
Description: Spirometry measurements were conducted in accordance with the current ATS/ERS 2005 guidelines.
Time Frame: 0 to 4hr
Population: all subjects who received at least one dose of the study medication and have at least one post baseline efficacy measurement were included in the efficacy population. . A subject received more than one treatment type throughout the study.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Glycopyrrolate Inhalation Solution 25mg | Glycopyrrolate Inhalation Solution 75mg | Glycopyrrolate Inhalation Solution 200mg | Glycopyrrolate Inhalation Solution 200mg Jet | Glycopyrrolate Inhalation Solution 500mg | Glycopyrrolate Inhalation Solution1000mg | Placebo 0.5 mL
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6
percent change | 17.12 (9.07) | 15.60 (4.20) | 22.98 (4.99) | 19.28 (13.10) | 11.47 (6.86) | 16.87 (6.83) | 6.80 (2.91)

12. Secondary Outcome: Peak FEV1 (Change From Baseline )
Description: Spirometry measurements were conducted in accordance with the current ATS/ERS 2005 guidelines.
Time Frame: 0 to 4hr
Population: All subjects who received at least one dose of study medication and have at least one post baseline efficacy measurement were included in the efficacy population.. A subject received more than one treatment type throughout the study.
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Glycopyrrolate Inhalation Solution 25mg | Glycopyrrolate Inhalation Solution 75mg | Glycopyrrolate Inhalation Solution 200mg | Glycopyrrolate Inhalation Solution 200mg Jet | Glycopyrrolate Inhalation Solution 500mg | Glycopyrrolate Inhalation Solution1000mg | Placebo 0.5 mL
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6
liters | 0.212 (0.086) | 0.255 (0.068) | 0.303 (0.055) | 0.233 (0.144) | 0.177 (0.061) | 0.283 (0.069) | 0.120 (0.057)

13. Secondary Outcome: FEV1 AUC0-24 Area Under the FEV1 Over Time Curve (Change From Baseline)
Description: Spirometry measurements were conducted in accordance with the current ATS/ERS 2005 guidelines.
Time Frame: 0 to 24hr post dose
Population: All subjects who received at least one dose of study medication and have at least one post baselineefficacy measurement were included in the efficacy population. A subject received more than one treatment type throughout the study.
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Glycopyrrolate Inhalation Solution 25mg | Glycopyrrolate Inhalation Solution 75mg | Glycopyrrolate Inhalation Solution 200mg | Glycopyrrolate Inhalation Solution 200mg Jet | Glycopyrrolate Inhalation Solution 500mg | Glycopyrrolate Inhalation Solution1000mg | Placebo 0.5 mL
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6
liters | 1.59 (3.27) | 3.10 (2.27) | 3.19 (1.14) | 1.35 (2.74) | 1.53 (2.05) | 3.08 (1.47) | -0.11 (1.89)

14. Secondary Outcome: Cmax Maximum Observed Plasma Concentration
Description: Pk parameters are calculated from glycopyrrolate plasma concentration analysed from serial blood samples collected between 0 and 12 hr
Time Frame: 0 to 12 hours post dose
Population: All subjects who received at least one dose of study medication and who have sufficient blood samples taken to obtain a plasma concentration by time profile were included in the PK . A subject received more than one treatment type throughout the study.
  analysis.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Glycopyrrolate Inhalation Solution 200mg | Glycopyrrolate Inhalation Solution 200mg Jet | Glycopyrrolate Inhalation Solution 500mg | Glycopyrrolate Inhalation Solution1000mg
Number analyzed (Participants) | 6 | 6 | 6 | 6
pg/mL | 177.242 (61.469) | 75.530 (64.950) | 749.872 (219.696) | 1534.057 (442.581)

15. Secondary Outcome: Tmax Time to Maximum Observed Plasma Concentration
Description: as for outcome 14
Time Frame: 0 to 12 hours post dose
Population: All subjects who received at least one dose of study medication and who have sufficient blood samples taken to obtain a plasma concentration by time profile were included in the PK analysis. A subject received more than one treatment type throughout the study.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Glycopyrrolate Inhalation Solution 200mg | Glycopyrrolate Inhalation Solution 200mg Jet | Glycopyrrolate Inhalation Solution 500mg | Glycopyrrolate Inhalation Solution1000mg
Number analyzed (Participants) | 6 | 6 | 6 | 6
hours | .025 (0.088) | 0.08 (0.088) | 0.25 (0.069) | 0.17 (0.093)

16. Secondary Outcome: AUC0-t Area Under the Plasma Concentration-time Curve From Time Zero to the Last Quantifiable Concentration
Description: as for outcome 14
Time Frame: 0 to 12 hourr post dose
Population: All subjects who received at least one dose of study medication and who have sufficient blood samples taken to obtain a plasma concentration by time profile were included in the PK analysis.A subject received more than one treatment type throughout the study.
Measure: Mean (Standard Deviation); unit: pg*h/mL
Arm/Group | Glycopyrrolate Inhalation Solution 200mg | Glycopyrrolate Inhalation Solution 200mg Jet | Glycopyrrolate Inhalation Solution 500mg | Glycopyrrolate Inhalation Solution1000mg
Number analyzed (Participants) | 6 | 6 | 6 | 6
pg*h/mL | 429.335 (192.699) | 26.176 (16.170) | 2014.276 (609.911) | 4084.763 (827.225)

17. Secondary Outcome: AUC0-inf Area Under the Plasma Concentration-time Curve From Time Zero to Infinity
Description: as for outcome 14
Time Frame: 0 to 12 hours post dose
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: pg*h/mL
Arm/Group | Glycopyrrolate Inhalation Solution 200mg | Glycopyrrolate Inhalation Solution 200mg Jet | Glycopyrrolate Inhalation Solution 500mg | Glycopyrrolate Inhalation Solution1000mg
Number analyzed (Participants) | 6 | 6 | 6 | 6
pg*h/mL | 563.416 (235.418) | 65.013 (16.750) | 2491.803 (736.426) | 5271.099 (1096.862)

18. Secondary Outcome: t1/2 Plasma Half-life
Description: as for outcome 14
Time Frame: 0 to 12 hours post-dose
Population: Subjects who received at least one dose of study medication and have sufficient blood samples taken to obtain a plasma concentration by time profile were included in the PK analysis.Subject received more than one treatment type throughout the study
  samples taken to obtain a plasma concentration by time profile were included in the PK analysis.
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Glycopyrrolate Inhalation Solution 200mg | Glycopyrrolate Inhalation Solution 200mg Jet | Glycopyrrolate Inhalation Solution 500mg | Glycopyrrolate Inhalation Solution1000mg
Number analyzed (Participants) | 6 | 6 | 6 | 6
hour | 2.947 (1.996) | 0.778 (0.465) | 6.298 (1.450) | 7.573 (1.031)

ADVERSE EVENTS:
Time Frame: 0-47 days
Description: AE's are defined as existing conditions which worsen or events which occur during the course of the clinical trial after treatment
Groups:
- Glycopyrrolate Inhalation Solution 25 μg: Glycopyrrolate Inhalation Solution 25 μg via eFlow nebulizer, once daily
  Glycopyrrolate Inhalation Solution 25mg: 25 μg oral inhalation via eFlow Nebulizer, once daily
- Glycopyrrolate Inhalation Solution75μg: Glycopyrrolate Inhalation Solution 75 μg via eFlow nebulizer, once daily
  Glycopyrrolate Inhalation Solution 75 μg via eFlow nebulizer, once daily
- Glycopyrrolate Inhalation Solution 200 μg: Glycopyrrolate Inhalation Solution 200 μg via eFlow nebulizer, once daily
  Glycopyrrolate Inhalation Solution 200 μg via eFlow nebulizer, once daily
- Glycopyrrolate Inhalation Solution 200μg Jet Nebulizer,: Glycopyrrolate Inhalation Solution 200μg Jet Nebulizer ,once daily
  Glycopyrrolate Inhalation Solution 200μg Jet Nebulizer, once daily
- Glycopyrrolate Inhalation Solution 500μg: Glycopyrrolate Inhalation Solution 500μg eFlow Nebulizer, once daily
  Glycopyrrolate Inhalation Solution 500μg eFlow Nebulizer, once daily
- Glycopyrrolate Inhalation Solution1000mg: Glycopyrrolate Inhalation Solution1000mg via eFlow nebulizer, once daily
  Glycopyrrolate Inhalation Solution1000mg via eFlow nebulizer, once daily
- Placebo: Placebo
  Placebo
Arm/Group | Glycopyrrolate Inhalation Solution 25 μg | Glycopyrrolate Inhalation Solution75μg | Glycopyrrolate Inhalation Solution 200 μg | Glycopyrrolate Inhalation Solution 200μg Jet Nebulizer, | Glycopyrrolate Inhalation Solution 500μg | Glycopyrrolate Inhalation Solution1000mg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 2/6 | 2/6 | 4/6 | 2/6 | 0/6 | 2/6 | 1/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Glycopyrrolate Inhalation Solution 25 μg (N=6) | Glycopyrrolate Inhalation Solution75μg (N=6) | Glycopyrrolate Inhalation Solution 200 μg (N=6) | Glycopyrrolate Inhalation Solution 200μg Jet Nebulizer, (N=6) | Glycopyrrolate Inhalation Solution 500μg (N=6) | Glycopyrrolate Inhalation Solution1000mg (N=6) | Placebo (N=6)
catheter site related reaction (General disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 2 (2) | 1 (1)
nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
headache (Nervous system disorders) | 1 (1) | 1 (2) | 3 (4) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In the event the Study is part of a multi-center study, the first publication of the results of the Study shall be made in conjunction with the results of other participating study sites as a multi-center publication; provided however, if a multi-center publication is not forthcoming within twenty-four (24) months following completion of the Study at all sites, Institution and Investigator shall be free to publish.